CLINICAL TRIAL: NCT02170896
Title: Bioavailability of BIBR 953 ZW After 50 mg of BIBR 1048 MS (Oral Prodrug of BIBR 953) in 4 Experimental Formulations Relative to Drinking Solution of BIBR 1048 MS, Each Treatment Given Bid Over 3 Days, in Healthy Subjects. Intraindividual Comparison (5-way Crossover), Randomised, Open. For Each of the 5 Treatments, Investigation of 2 Conditions: With and Without Pantoprazole (Intraindividual, Open Comparison).
Brief Title: Bioavailability of BIBR 963 ZW After 50 mg of BIBR 1048 MS With and Without of Pantoprazole in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.31
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Fumigant 93; Pantoprazole

ARMS (8):
- Period 1: BIBR1048 MS Capsule A+Pantoprazole (Experimental)
  Interventions: Drug: BIBR 1048 MS Capsule A; Drug: Pantoprazole
- Period 1: BIBR1048 MS Capsule B+Pantoprazole (Experimental)
  Interventions: Drug: BIBR 1048 MS Capsule B; Drug: Pantoprazole
- Period 1: BIBR1048 MS Capsule C+Pantoprazole (Experimental)
  Interventions: Drug: BIBR 1048 MS Capsule C; Drug: Pantoprazole
- Period 1: BIBR1048 MS Capsule D+Pantoprazole (Experimental)
  Interventions: Drug: BIBR 1048 MS Capsule D; Drug: Pantoprazole
- Period 1: BIBR1048 MS solution+Pantoprazole (Active Comparator)
  Interventions: Drug: BIBR 1048 MS tartaric acid solution; Drug: Pantoprazole
- Period 2: BIBR1048 MS Capsule C (Experimental)
  Interventions: Drug: BIBR 1048 MS Capsule C
- Period 2: BIBR1048 MS Capsule D (Experimental)
  Interventions: Drug: BIBR 1048 MS Capsule D
- Period 2: BIBR1048 MS solution (Active Comparator)
  Interventions: Drug: BIBR 1048 MS tartaric acid solution

INTERVENTIONS:
Drug: BIBR 1048 MS Capsule A
  Arms: Period 1: BIBR1048 MS Capsule A+Pantoprazole
Drug: BIBR 1048 MS Capsule B
  Arms: Period 1: BIBR1048 MS Capsule B+Pantoprazole
Drug: BIBR 1048 MS Capsule C
  Arms: Period 1: BIBR1048 MS Capsule C+Pantoprazole; Period 2: BIBR1048 MS Capsule C
Drug: BIBR 1048 MS Capsule D
  Arms: Period 1: BIBR1048 MS Capsule D+Pantoprazole; Period 2: BIBR1048 MS Capsule D
Drug: BIBR 1048 MS tartaric acid solution
  Arms: Period 1: BIBR1048 MS solution+Pantoprazole; Period 2: BIBR1048 MS solution
Drug: Pantoprazole
  Arms: Period 1: BIBR1048 MS Capsule A+Pantoprazole; Period 1: BIBR1048 MS Capsule B+Pantoprazole; Period 1: BIBR1048 MS Capsule C+Pantoprazole; Period 1: BIBR1048 MS Capsule D+Pantoprazole; Period 1: BIBR1048 MS solution+Pantoprazole

SUMMARY:
To assess the amount of BIBR 953 ZW in urine of 50 mg of BIBR 1048 bid over three days each administered as four experimental capsule formulations relative to drinking solution with and without coadministration of 40 mg pantoprazole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with GCP (Good Clinical Practice) and local legislation
* Age >= 18 and <= 55 years
* Body Mass Index (BMI) >= 18.5 and <= 29.9 kg/m²

Exclusion Criteria:

* Any finding at the medical examination (including blood pressure, pulse rate and ECG (electrocardiogram)) deviation from normal and of clinical relevance
* History of or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of relevant orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* History of any bleeding disorder including prolonged or habitual bleeding
* History of other hematologic disease
* History of cerebral bleeding (e.g. after a car accident)
* History of commotio cerebri
* Intake of drug with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs that might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familial bleeding disorder
* Thrombocytes < 150000/µl

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2001-10; Primary Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Ae 0-12h: amount of drug (total BIBR 953 ZW) excreted into urine during all individual dosing intervals | up to 3 days after each administration
Area under the concentration time course at steady state (AUCss) | 0.5, 1, 1.5, 2, 4, 6, 8 and 12 hours after study drug administration on day 3 of period 2

SECONDARY OUTCOMES:
Occurence of adverse events | up to 40 days
Maximum plasma concentration at steady state (Cmax,ss) | 0.5, 1, 1.5, 2, 4, 6, 8 and 12 hours after study drug administration on day 3 of period 2
Time at which maximum plasma concentration occurs after dosing during steady state (tmax,ss) | 0.5, 1, 1.5, 2, 4, 6, 8 and 12 hours after study drug administration on day 3 of period 2